CLINICAL TRIAL: NCT01228565
Title: Placebo Controlled Randomized Trial of OTD70DERM® in Radio-dermatitis Induced by Radiotherapy-Erbitux®
Brief Title: Trial of OTD70DERM® in Radio-dermatitis Induced by Radiotherapy-Erbitux®
Acronym: GORTEC 2009-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GORTEC 2009-01
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Head and Neck Carcinoma
Keywords: Head and neck carcinoma treated by radiotherapy plus erbitux
MeSH Terms: interventions — Radiotherapy; Cetuximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Radiotherapy+Erbitux+Placebo
  Interventions: Other: Radiotherapy + Erbitux® + placebo
- OTD70DERM (Experimental): Radiotherapy+Erbitux+OTD70DERM®
  Interventions: Other: Radiotherapy+Erbitux+OTD70DERM

INTERVENTIONS:
Other: Radiotherapy + Erbitux® + placebo — 3D radiotherapy 70 Gy / 7 weeks (no IRMT); Erbitux once a week, 1 week before radiotherapy and during radiotherapy ; Placebo local application, once a day, every day during the radiotherapy
  Arms: Placebo
Other: Radiotherapy+Erbitux+OTD70DERM — 3D radiotherapy 70 Gy / 7 weeks (no IRMT); Erbitux once a week, 1 week before radiotherapy and during radiotherapy ; OTD70DERM local application, once a day, every day during the radiotherapy
  Arms: OTD70DERM

SUMMARY:
The aim of this randomized trial is to compare the rate of radio-dermatitis grade 2+ (NCI-CTC V3.0) in patients receiving radiotherapy+Erbitux+placebo versus in patients receiving radiotherapy+Erbitux+OTD70DERM® for the treatment of head and neck carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck carcinoma treated by radiotherapy (70Gy) plus Erbitux

Exclusion Criteria:

* IMRT; Concomitant chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Radio-dermatitis grade 2, 3, 4 (NCI-CTC V3) | 3 months
  Radio-dermatitis grade 2, 3, 4 (according to the NCI-CTC V3. Radio-dermatitis will be evaluated twice a week during radiotherapy and at M1, M2 and M3 after end of treatment.

SECONDARY OUTCOMES:
Quality of life | 3 months
  Quality of life by the Dermatology Life Quality Index (DLQI)

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHI Creteil, Créteil
  - Centre de Forcilles, Ferolles Attily
  - CLCC Nantes, Nantes
  - CHU Pitie Salpetriere, Paris
  - Institut Gustave Roussy, Villejuif